CLINICAL TRIAL: NCT01941589
Title: Combination Corticosteroids + 5-aminosalicylic Acids Compared to Corticosteroids Alone in the Treatment of Moderate-severe Active Ulcerative Colitis.
Brief Title: Corticosteroids+5-aminosalicylic Acid Compared to Corticosteroids in the Treatment of Moderate-severe Ulcerative Colitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofir Harnoy MD, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-13-0401-OH-CTIL
Record Dates: First submitted 2013-08-30; First posted 2013-09-13 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; Hydrocortisone; hydrocortisone hemisuccinate; Methylprednisolone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- present 5-ASA arm 1 (Active Comparator): oral 5-ASA+/-topical 5-ASA+IV corticosteroids / PO Methylprednisolone
  Interventions: Drug: oral 5-ASA+/-topical 5-ASA+IV corticosteroids / PO Methylprednisolone
- 5-ASA naive arm 1 (Active Comparator): oral 5-ASA+/-topical 5-ASA+IV corticosteroids / PO Methylprednisolone
  Interventions: Drug: oral 5-ASA+/-topical 5-ASA+IV corticosteroids / PO Methylprednisolone
- present 5-ASA arm 2 (Active Comparator): IV corticosteroids only / PO Methylprednisolone
  Interventions: Drug: corticosteroids only
- 5-ASA naive arm 2 (Active Comparator): IV corticosteroids only / PO Methylprednisolone
  Interventions: Drug: corticosteroids only

INTERVENTIONS:
Drug: oral 5-ASA+/-topical 5-ASA+IV corticosteroids / PO Methylprednisolone — maximal oral 5-ASA+/-topical 5-ASA+IV corticosteroids
  Other Names: rafassal; pentasa; asacol; hydrocortisone; solu-cortef; methylprednisolone
  Arms: 5-ASA naive arm 1; present 5-ASA arm 1
Drug: corticosteroids only — IV corticosteroids only
  Other Names: hydrocortisone; solu-cortef; methylprednisolone
  Arms: 5-ASA naive arm 2; present 5-ASA arm 2

SUMMARY:
The role of steroids in the treatment of ulcerative Colitis (UC) is well established, and recommended by professional societies. However, there are no data investigating whether the addition and/or continuation of 5-aminosalicylic agents as combination therapy with systemic corticosteroids is superior to corticosteroids alone in patients with moderate-severe active UC. Thus, in practical terms, the decision regarding 5-aminosalicylic (to add or continue), on top of steroids treatment, is taken on an arbitrary basis. The aim of this study is to compare the efficacy of steroids alone Vs combination of steroids + 5-aminosalicylic in the treatment of moderate-severe UC exacerbation.

DETAILED DESCRIPTION:
he role of steroids in the treatment of ulcerative Colitis (UC) is well established, and recommended by professional societies. However, there are no data investigating whether the addition and/or continuation of 5-aminosalicylic agents as combination therapy with systemic corticosteroids is superior to corticosteroids alone in patients with moderate-severe active UC. Thus, in practical terms, the decision regarding 5-aminosalicylic (to add or continue), on top of steroids treatment, is taken on an arbitrary basis. The aim of this study is to compare the efficacy of steroids alone Vs combination of steroids + 5-aminosalicylic in the treatment of moderate-severe UC exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* UC known and diagnosed by established clinical-endoscopic and histological criteria or newly-diagnosed UC, based on clinical and endoscopic findings, and about to start treatment with corticosteroids.
* current hospitalization with severe Ulcerative Colitis exacerbation as defined by a Lichtiger score of >10
* age >18
* if taking thiopurines, the dose must be stable for 2 months prior to admission

Exclusion Criteria:

* pregnant women
* allergy/unable to take study medications
* active infection
* severe renal/liver/cardiorespiratory condition
* toxic megacolon or signs of imminent colectomy
* treatment with an anti-tumor necrosis factor in 3 months prior to admission
* prior treatment with cyclosporin or tacrolimus
* alcohol dependancy
* unwilling/ unable to give an informed consent
* participation in clinical trials in the last 2 months prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-09; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
percentage of patients who respond to the treatment | day 7

SECONDARY OUTCOMES:
the percentage of patients in need of a rescue medication | day 5, 7
colectomy rate | 1 month, 3 months post randomization

OTHER OUTCOMES:
duration of hospitalization | 3-90

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Har-Noy, MD, Principal Investigator — Sheba Medical Center, Tel-Hashomer, ISRAEL 52621
Locations (10):
- China (2):
  - 6th affiliated hospital of Sun yat-sen university, Guangzhou
  - Department of Gastroenterology and Hepatology,The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
- Service de Gastrologie-Entérologie-Hépatologie, Centre Hospitalier Universitaire de Saint-Étienne, Saint-Etienne, France
- Greece (2):
  - Department of Gastroenterology Venizeleio General Hospital, Leoforos Knosou, Heraklion
  - Department of Gastroenterology, University Hospital & Medical School of Ionnina, Ioannina
- Israel (2):
  - Gastroenterology department, Soroka medical center, Beersheba
  - Sheba Medical Center, Tel Litwinsky
- Università di Roma Sapienza, Rome, Italy
- Zvezdara University Clinical Center, Gastroenterology Department, Belgrade, Serbia
- nstitute of Gastroenterology and Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ben-Horin S, Har-Noy O, Katsanos KH, Roblin X, Chen M, Gao X, Schwartz D, Cheon JH, Cesarini M, Bojic D, Protic M, Theodoropoulou A, Abu-Kaf H, Engel T, Tang J, Veyrard P, Lin X, Mao R, Christodoulou D, Karmiris K, Knezevic-Ivanovski T; ComboMesa investigators. Corticosteroids and Mesalamine Versus Corticosteroids for Acute Severe Ulcerative Colitis: A Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2868-2875.e1. doi: 10.1016/j.cgh.2022.02.055. Epub 2022 Mar 8. PMID 35272029